CLINICAL TRIAL: NCT05824351
Title: Team LowCostomy: Dedicated Toward Creating a High-quality, Low-cost Colostomy Appliance for Those in Sub-Saharan Africa and Other Low Resource Settings.
Brief Title: LowCostomy: Dedicated Toward Creating a High-quality, Low-cost Colostomy Appliance for Those in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: VentureWell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00111440
Record Dates: First submitted 2023-03-20; First posted 2023-04-21 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Abdominal Site; Colostomy Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Tanzanian beeswax-pine adhesive (Experimental): Each study subject will be tested with a thin ring of adhesive in the form of a Tanzanian beeswax-pine resin formula.
  Interventions: Device: Tanzanian beeswax-pine resin
- Domestic beeswax-pine adhesive (Active Comparator): Each study subject will be tested with a thin ring of adhesive in the form of a domestic beeswax-pine resin formula.
  Interventions: Device: Domestic beeswax-pine resin
- Control (Active Comparator): Each study subject will be tested with a thin ring of adhesive in the form of Hollister's AdaptTM Barrier Rings.
  Interventions: Device: Hollister's AdaptTM Barrier Rings

INTERVENTIONS:
Device: Tanzanian beeswax-pine resin — Thin ring of adhesive in the form of a Tanzanian beeswax-pine resin formula.
  Arms: Tanzanian beeswax-pine adhesive
Device: Domestic beeswax-pine resin — Thin ring of adhesive in the form of a domestic beeswax-pine resin formula.
  Arms: Domestic beeswax-pine adhesive
Device: Hollister's AdaptTM Barrier Rings — Thin ring of adhesive in the form of Hollister's AdaptTM Barrier Rings.
  Arms: Control

SUMMARY:
The purpose of this study is to examine the safety of the LowCostomy appliance's peristomal adhesive interface composed of a mix of beeswax and pine resin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with age +/>18 years
* Recruited from Duke University
* Local community members

Exclusion Criteria:

* Any pre-existing skin conditions
* Skin allergies to tegaderm or other adhesive products contained within the study and control rings

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Barto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Denter, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control: Each study subject will be tested with thin rings of three types of adhesive.
  Tanzanian beeswax-pine resin: Thin ring of adhesive in the form of a Tanzanian beeswax-pine resin formula.
  Domestic beeswax-pine resin: Thin ring of adhesive in the form of a domestic beeswax-pine resin formula.
  Control: Thin ring of adhesive in the form of Hollister's AdaptTM Barrier Rings.
Period: Overall Study
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Started | 50
Completed | 44
Not Completed | 6
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Skin Irritation as Measured by Draize Score for Erythema and Edema
Description: The Draize score (for each erythema and edema) has a range of 0 to 4, where a higher score indicated greater irritation. Individual scores below 3 were classified as not severe.
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 9 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tanzanian Beeswax-pine Adhesive | Domestic Beeswax-pine Adhesive | Control
Number analyzed (Participants) | 35 | 35 | 35
score on a scale
  Edema | 0.86 (0.28) | 0.03 (0.17) | 0 (0)
  Erythema | 0.38 (0.65) | 0.15 (0.50) | 0.44 (0.66)
Statistical Analysis 1: Comparison: Domestic Beeswax-pine Adhesive vs Control; Draize scores for erythema/eschar and edema were summed for analysis (range of 0 to 8, where a higher score indicated greater irritation); Test type: Equivalence — Equivalence is defined as an average difference of < or = 2; p < 0.0001, t-test, 1 sided; One-sided lower t-test; Mean of paired differences = -0.2571, Standard Deviation 0.70
Statistical Analysis 2: Comparison: Tanzanian Beeswax-pine Adhesive vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Equivalence is defined as an average difference of < or = 2; p = 0.0003, t-test, 1 sided; One-sided upper t-test; Mean of paired differences = 0.0294, Standard Deviation 0.79

2. Primary Outcome: Skin Irritation as Measured by the 5-D (5-dimension) Itch Scale
Description: The 5-D Itch Scale is a questionnaire consisting of 5 items used specifically to measure the course of itch by asking for the degree, duration, disability and distribution of the itching. The score ranges from 5 to 25, where a higher score indicates greater itching.
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Data not collected.
Arm/Group | Tanzanian Beeswax-pine Adhesive | Domestic Beeswax-pine Adhesive | Control
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Skin Irritation as Measured by Survey: "During the Last Week, How Many Hours a Day Have You Been Itching?"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Less than 6hrs/day" | 40
  "6-12 hrs/day" | 2

4. Primary Outcome: Skin Irritation as Measured by Survey: "Please Rate the Intensity of Your Itching Over the Past Two Weeks"
Time Frame: Assessed daily up to 14 days, day 14 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Not Present" | 17
  "Mild" | 20
  "Moderate" | 5

5. Primary Outcome: Skin Irritation as Measured by Survey: "Over the Past Week, Has Your Itching Progressively Gotten Better or Worse?"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Getting worse" | 7
  "Unchanged" | 10
  "Little bit better, but still present" | 4
  "Much better, but still present" | 2
  "Completely resolved" | 2
  "Not relevant/applicable" | 17

6. Primary Outcome: Skin Irritation as Measured by Survey: "Rate the Impact of Your Itching (if Any) on SLEEP Over the Last Week"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Never affects sleep" | 37
  "Occasional delays in falling asleep" | 5

7. Primary Outcome: Skin Irritation as Measured by Survey: "Rate the Impact of Your Itching (if Any) on LEISURE/SOCIAL ACTIVITIES Over the Last Week"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Never affects this activity" | 23
  "Rarely affects this activity" | 1
  "Occasionally affects this activity" | 2
  "Not relevant/applicable" | 16

8. Primary Outcome: Skin Irritation as Measured by Survey: "Rate the Impact of Your Itching (if Any) on HOUSEWORK/ERRANDS Over the Last Week"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Never affects this activity" | 24
  "Rarely affects this activity" | 2
  "Occasionally affects this activity" | 0
  "Not relevant/applicable" | 16

9. Primary Outcome: Skin Irritation as Measured by Survey: "Rate the Impact of Your Itching (if Any) on WORK/SCHOOL Over the Last Week"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Never affects this activity" | 24
  "Rarely affects this activity" | 2
  "Occasionally affects this activity" | 0
  "Not relevant/applicable" | 16

10. Primary Outcome: Skin Irritation as Measured by Survey: "Mark Whether the Itching (if Any) Spread to the Following Parts of Your Body"
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data not collected on 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 42
Participants
  "Broader Abdomen" | 2
  "Unchecked" | 1
  "Not relevant/applicable" | 39

11. Secondary Outcome: Number of Participants With Adverse Side Effects Such as Redness, Rash, Skin Irritation, and Infection
Time Frame: Assessed daily up to 7 days, day 7 reported
Population: Each participant received all three types of adhesive. Data were collected on the whole participant level for the reported adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 50
Participants | 6

12. Secondary Outcome: Overall Well-being as Measured by Daily Survey
Description: Number of participants who responded "yes" to the question, "Have you had any major discomfort/irritation/redness/swelling caused any of the three samples?"
Time Frame: Daily, days 1-7
Population: Participants with data collected at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 44
Participants
  Day 1 | 0
  Day 2 | 0
  Day 3 | 0
  Day 4 | 0
  Day 5 | 1
  Day 6 | 0
  Day 7: number analyzed (Participants) | 42
  Day 7 | 2

13. Secondary Outcome: Overall Well-being as Measured by Daily Survey
Description: Number of participants who responded "yes" to the question, "Were you able to successfully remove and reattach all three samples + Tegaderm (the clear adhesive) today?"
Time Frame: Daily, days 1-6
Population: Participants with data collected at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 44
Participants
  Day 1 | 44
  Day 2 | 44
  Day 3 | 43
  Day 4 | 42
  Day 5 | 42
  Day 6 | 44

14. Secondary Outcome: Overall Well-being as Measured by Daily Survey
Description: Number of participants who responded "yes" to the question, "Were any of your samples removed for longer than 20 minutes at any point today?"
Time Frame: Daily, days 1-7
Population: Participants with data collected at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
Number analyzed (Participants) | 44
Participants
  Day 1 | 2
  Day 2 | 1
  Day 3 | 0
  Day 4 | 2
  Day 5 | 2
  Day 6 | 1
  Day 7: number analyzed (Participants) | 42
  Day 7 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: Each participant received all three types of adhesive. Data were collected on the whole participant level for the reported adverse events data.
Arm/Group | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanzanian Beeswax-pine Adhesive, Domestic Beeswax-pine Adhesive, and Control (N=50)
Skin redness/irritation (Skin and subcutaneous tissue disorders) | 6 — Expected adverse event due to the adhesive bandage used, not the study products.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05824351/Prot_001.pdf